CLINICAL TRIAL: NCT07370051
Title: Effect of Topical Oxygen and LED Light Therapy on Nipple Crack: A Randomized Controlled Trial
Brief Title: Effect of Topical Oxygen and LED Light Therapy on Nipple Crack
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Elif Dogan, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025/xxx
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Breastfeeding; Newborn Infant; Midwifery; Breast
MeSH Terms: conditions — Breast Feeding | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Topical oxygen therapy group (Experimental)
  Interventions: Procedure: Topical oxygen therapy
- LED light therapy group (Experimental)
  Interventions: Device: LED light therapy
- Control group (No Intervention)

INTERVENTIONS:
Procedure: Topical oxygen therapy — Topical oxygen will be applied directly to the nipple crack using an oxygen mask. The oxygen mask will be washed and dried before and after use. The mask, which is specific to the individual, will be stored in a transparent, sealed plastic bag until it is reused.
  In the literature, free-flow oxygen applications are frequently administered at a rate of 5-15 liters/min for 10-180 minutes.
  The size of the nipple fissure is smaller than most wound types reported in the literature. Therefore, considering the wound size and the need to avoid long application times that would compromise maternal comfort, the therapeutic dose was adjusted accordingly. In line with this, after consulting a surgical specialist, it was planned to administer one session at a flow rate of 10 liters per minute for 20 minutes. The determined application parameters will be tested in a pilot study.
  Arms: Topical oxygen therapy group
Device: LED light therapy — An LED light device based on the photobiomodulation principle, commonly used in clinical dermatology applications, will be used in LED light therapy. The LED light will be applied directly to the nipple crack. The device is recommended to be used at a distance of 3 inches (~8 cm). The application time was determined by calculating the formulation used in similar studies in the literature: Time (sec) = Energy dose (J/cm²) ÷ Light intensity (W/cm²). Thus, the ideal duration for the device to be used was determined to be 300 seconds (5 minutes), as 15.3 J/cm² ÷ 0.051 W/cm². LED light will only be applied to Group B and a total of three times (day 0, day 3, day 7).
  Arms: LED light therapy group

SUMMARY:
The World Health Organization and UNICEF define the protection and support of breastfeeding as one of the key determinants of maternal and newborn health. Nipple cracks are common in the postpartum period and cause breastfeeding problems. If not addressed early, they can lead to interrupted or complete cessation of breastfeeding. It is important to develop methods for effective, safe, and mother-friendly care of nipple cracks. Various care approaches, such as lanolin, natural products, and hydrogels, have been described in the literature. However, evidence for non-invasive agents that support wound healing at the cellular level is limited. Evidence for LED light application is limited, and there is no evidence regarding the effect of topical oxygen application on nipple cracks.

This project is designed as a randomized controlled trial to investigate the effect of topical oxygen and LED light therapy applied to nipple cracks on wound healing, pain, and breastfeeding success. The study will be conducted at the Lactation Unit of Istanbul Haseki Training and Research Hospital, Ministry of Health, between March and December 2026. The sample size was calculated using the G*Power program; with an effect size of 0.20, a significance level of 5%, and a power of 80%, a total of 51 mothers will be included in the study. Participants will be divided into three groups using the block randomization method: Topical Oxygen (n=17), LED Light Therapy (n=17), and Control (n=17). Standard breastfeeding counseling will be provided to all groups. In addition to the intervention groups, topical oxygen will be applied at a flow rate of 10 liters per minute for 20 minutes; LED light therapy will be applied at 630 nm red and 850 nm infrared wavelengths, at an energy dose of 15.3 J/cm², for 5 minutes. Interventions will be performed on days 0, 3, and 7. Data will be collected using a personal information form, wound size measurement, Nipple Trauma Score, Visual Analog Scale, and LATCH score. The validity and reliability of the Nipple Trauma Score in Turkish will be assessed within the scope of the project.

To reduce measurement and analysis bias, support will be obtained from an independent observer and a statistician.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-40,
* Those who gave birth at term (37-42 weeks),
* Those whose baby was 0-28 days old at the first visit,
* Those diagnosed with nipple fissures,
* Breastfeeding their baby,
* Those who have had a single birth,
* Those without a diagnosis of psychiatric illness and who are not taking related medication.

Exclusion Criteria:

* Those with infection, mastitis, abscess, etc. accompanying nipple injury,
* Those who have started medical treatment for nipple injury,
* Those who are unable to continue breastfeeding,
* Those who feed their baby by expressing breast milk,
* Those who show any adverse reaction to photosensitivity or exposure to sunlight.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Eligibility is limited based on biological sex, as the study includes postpartum individuals who have given birth and are breastfeeding.
Enrollment: 51 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Nipple Trauma Severity | Day 1 (pre- and post-intervention), Day 3 (post-intervention), and Day 7 (post-intervention)
  Nipple trauma severity will be assessed using the Nipple Trauma Score (NTS), which evaluates breastfeeding-related nipple tissue damage based on objective observational criteria. The scale categorizes nipple changes into six severity levels scored from 0 to 5, with higher scores indicating more severe nipple trauma. The Turkish version of the scale will be developed and used in this study.
Nipple Pain Intensity | Day 1 (pre- and post-intervention), Day 3 (post-intervention), and Day 7 (post-intervention)
  Nipple pain intensity will be measured using the Visual Analog Scale (VAS), a 10-cm subjective pain scale ranging from 0 (no pain) to 10 (unbearable pain). Participants will indicate the intensity of pain related to nipple trauma by marking the scale, with higher scores reflecting greater pain severity.

SECONDARY OUTCOMES:
Breastfeeding Effectiveness (LATCH Score) | Day 1 (pre- and post-intervention), Day 3 (pre-intervention), and Day 7 (pre-intervention)
  Breastfeeding effectiveness will be evaluated using the LATCH Breastfeeding Assessment Tool, which assesses latch, audible swallowing, nipple type, maternal comfort, and need for assistance. Each component is scored from 0 to 2, yielding a total score range of 0 to 10, with higher scores indicating more effective breastfeeding.
Infant Weight Change | Day 1 (pre-intervention), Day 3 (pre-intervention), and Day 7 (pre-intervention)
  Infant weight will be measured using a calibrated digital infant scale to assess changes in body weight over time. Weight measurements will be recorded in grams, and changes in infant weight will be used as an indicator of early feeding adequacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University - Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaves ME, Araujo AR, Santos SF, Pinotti M, Oliveira LS. LED phototherapy improves healing of nipple trauma: a pilot study. Photomed Laser Surg. 2012 Mar;30(3):172-8. doi: 10.1089/pho.2011.3119. Epub 2012 Jan 27. PMID 22283620
- [Background] Camargo BTS, Coca KP, Amir LH, Correa L, Aranha ACC, Marcacine KO, Abuchaim ESV, Abrao ACFV. The effect of a single irradiation of low-level laser on nipple pain in breastfeeding women: a randomized controlled trial. Lasers Med Sci. 2020 Feb;35(1):63-69. doi: 10.1007/s10103-019-02786-5. Epub 2019 Apr 27. PMID 31030379
- [Background] de Smet GHJ, Kroese LF, Menon AG, Jeekel J, van Pelt AWJ, Kleinrensink GJ, Lange JF. Oxygen therapies and their effects on wound healing. Wound Repair Regen. 2017 Aug;25(4):591-608. doi: 10.1111/wrr.12561. Epub 2017 Aug 7. PMID 28783878
- [Background] Sykorova M, Moffatt CJ, Stentiford N, Burian EA, Katsuhiro S, Wei Y. Topical oxygen therapy and singlet oxygen in wound healing: A scoping review. Int Wound J. 2024 Apr;21(4):e14846. doi: 10.1111/iwj.14846. PMID 38522472